CLINICAL TRIAL: NCT05952271
Title: Nationwide Retrospective Observational Study of Herpes Zoster Associated Hospital Admissions in Italy
Brief Title: Herpes Zoster Hospitalizations in Italy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of L'Aquila (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Antonella Mattei, Associate Professor, University of L'Aquila
Other Study IDs: 14112
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Herpes Zoster; Comorbidities and Coexisting Conditions
Keywords: Herpes Zoster; Vaccination; Hospitalizations; Comorbidities
MeSH Terms: conditions — Herpes Zoster | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hospitalization — Population of patients hospitalized for Herpes Zoster (ICD9-CM 053.xx)

SUMMARY:
In Italy, the 2017-2019 National Immunization Plan recommended specific vaccinations for the elderly, defined as those 65 years old and older, and at-risk adults with age 50+ (adults presenting cardiovascular, respiratory, or metabolic diseases, immunodepression, etc.). However, the coverage target set by the Plan (50% for Herpes Zoster vaccination in 2019) was not reached.

Providing additional data on the incidence of Herpes Zoster could improve the risks perception of the disease and the vaccination uptake. The present study will aim to describe a full picture of Herpes Zoster associated hospital admissions in Italy, focusing on co-morbidities which induce reduced varicella-zoster virus-specific cell-mediated immunity response. Furthermore, as varicella-zoster virus reactivation was reported in COVID-19-positive patients, a deepening on a possible relationship between the two infections will be investigated.

DETAILED DESCRIPTION:
Varicella (chickenpox) is a highly contagious illness sustained by an α Herpes virus called varicella-zoster virus (VZV). A replication phase in the penetration site is followed by a viremic phase when VZV spreads to skin and mucosae, leading to the typical rash and infection of sensory nerves in the epithelium, and then the reach of the sensory ganglia where it becomes latent. The reactivation of the latent virus, years or decades after primary infection, causes the typical clinical expression called Herpes Zoster (HZ) or shingles.

Post-herpetic neuralgia (PHN), an intractable pain in the dermatome affected by HZ, is the most common complication. It is estimated that it affects 10-20% of all patients with HZ aged ≥ 50 years and up to 30% of those aged ≥80 years. Management of PHN is not easy, but vaccination for prevention of PHN may be a strategic choice.

The most common complications of herpes zoster, other than PHN, often requiring hospitalization, include secondary bacterial infections, ophthalmic complications, cranial and peripheral nerve palsies, and segmental zoster paresis.

All authors agree that factors such as age, cell-mediated immunity (CMI) depression, intrauterine exposure to VZV and varicella occurring in early age (<18 months) are typically associated with HZ incidence. It further should be noted that age and CMI depression are strictly related since increasing age leads to CMI decrease. An increased incidence of hospitalization for HZ among patients aged >72 years (0.46/1000-person year), compared to those aged 15-44 years (0.03/1000-person year) was reported, suggesting that aging is also a risk factor for HZ requiring hospitalization. Besides age, HZ risk can be related to other co-morbidities, including diabetes, major depression or immunosuppressive therapies, that induce reduced VZV-specific CMI response. Immunosuppressed patients are within the high-risk group, with increasing morbidity and mortality associated with herpes zoster. Immunosuppression may be associated with malignancy (especially hematological), human immunodeficiency virus (HIV) infection or medications used for organ transplantation or autoimmune disease.

HZ incidence is similar all over the world and its trend is related to population age, with two thirds of the cases affecting subjects aged >50 years.

Among European adult population, the percentage of subjects estimated to be seropositive for anti-VZV antibodies is 95%: all of them are therefore potentially susceptible to develop HZ in their lifetime. In Italy, the annual incidence of HZ is 6.3/1000 person-years, with 73% of cases affecting adults.

Italy is one of the countries with the highest proportion of elderly people in its population, and yet data on the epidemiology of HZ and PHN are limited. As the immune system weakens with increasing age, many infectious diseases, such as HZ, are more severe and more closely associated with long-term consequences in the elderly than in younger people. With the growing aging population, a rise in the number of cases of HZ in the near future is expected; thus, this disease will become a public health issue. While awareness of childhood vaccination is well established, the prevention of infectious diseases in groups other than children is a challenging, yet fundamental, objective that public health systems should pursue in order to promote healthy aging.

In order to evaluate the epidemiological burden of HZ, hospital discharge records for HZ between 2011 and 2021, with or without complications, will be extracted from the national hospital discharge database (HDD).

The characteristics of hospitalizations will be described for the 18 years of age and older adults (2011-2021 years).

The characteristics of hospitalizations in 2020-21 will be described in patients with or without concomitant COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Hospital discharge records for Herpes Zoster infection in primary diagnosis age ≥18 years
* Hospital discharge records for Herpes Zoster infection in secondary diagnoses age ≥18 years

Exclusion Criteria:

* Hospital discharge records for Herpes Zoster infection in primary diagnosis age <18 years
* Hospital discharge records for Herpes Zoster infection in secondary diagnoses age <18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital discharge records for Herpes Zoster between 2011 and 2021, with or without complications, will be extracted from the national hospital discharge database (HDD).
  The characteristics of hospitalizations will be described for the 18 years of age and older adults (2011-2021 years).
  The characteristics of hospitalizations in 2020-21 will be described in patients with or without concomitant COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 72000 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Co-morbidities among Herpes Zoster hospitalizations | 2011-2021
  Rate of patients hospitalized for Herpes Zoster with co-morbidities

SECONDARY OUTCOMES:
Shingles annual hospitalization rates | 2011-2021
  Shingles annual hospitalization rates in the Italian adult population aged 18+
Shingles hospitalization rates by age classes | 2011-2021
  Shingles hospitalization rates by age classes:18-30; 31-40; 41-50; >50
Herpes Zoster and COVID-19 infection | 2020-2021
  Proportion of patients with HZ vs. patients with HZ and COVID-19 infection
Risk factors associated to deaths, a longer length of stay in hospital or the presence of zoster-complications among Herpes Zoster-related hospitalizations in the entire Italian general adult population | 2011-2021
  Incidence Rate Ratio (IRR) of deaths, longer length of stay in hospital or presence of zoster-complications among Herpes Zoster-related hospitalizations in the entire Italian general adult population

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Mattei, PhD, Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabutti G, Franco E, Bonanni P, Conversano M, Ferro A, Lazzari M, Maggi S, Rossi A, Scotti S, Vitale F, Volpi A, Greco D. Reducing the burden of Herpes Zoster in Italy. Hum Vaccin Immunother. 2015;11(1):101-7. doi: 10.4161/hv.34363. Epub 2014 Nov 1. PMID 25483522
- [Background] Grose C. Varicella vaccination of children in the United States: assessment after the first decade 1995-2005. J Clin Virol. 2005 Jun;33(2):89-95; discussion 96-8. doi: 10.1016/j.jcv.2005.02.003. PMID 15911422
- [Background] Gabutti G, Serenelli C, Cavallaro A, Ragni P. Herpes zoster associated hospital admissions in Italy: review of the hospital discharge forms. Int J Environ Res Public Health. 2009 Sep;6(9):2344-53. doi: 10.3390/ijerph6092344. Epub 2009 Sep 2. PMID 19826547
- [Background] Koshy E, Mengting L, Kumar H, Jianbo W. Epidemiology, treatment and prevention of herpes zoster: A comprehensive review. Indian J Dermatol Venereol Leprol. 2018 May-Jun;84(3):251-262. doi: 10.4103/ijdvl.IJDVL_1021_16. PMID 29516900
- [Background] Gialloreti LE, Merito M, Pezzotti P, Naldi L, Gatti A, Beillat M, Serradell L, di Marzo R, Volpi A. Epidemiology and economic burden of herpes zoster and post-herpetic neuralgia in Italy: a retrospective, population-based study. BMC Infect Dis. 2010 Aug 3;10:230. doi: 10.1186/1471-2334-10-230. PMID 20682044
- [Background] Stein AN, Britt H, Harrison C, Conway EL, Cunningham A, Macintyre CR. Herpes zoster burden of illness and health care resource utilisation in the Australian population aged 50 years and older. Vaccine. 2009 Jan 22;27(4):520-9. doi: 10.1016/j.vaccine.2008.11.012. Epub 2008 Nov 21. PMID 19027048
- [Background] Di Legami V, Gianino MM, Ciofi degli Atti M, Massari M, Migliardi A, Tomba GS, Zotti C; Zoster Study Group. Epidemiology and costs of herpes zoster: background data to estimate the impact of vaccination. Vaccine. 2007 Oct 23;25(43):7598-604. doi: 10.1016/j.vaccine.2007.07.049. Epub 2007 Aug 15. PMID 17889410
- [Background] Diez-Domingo J, Weinke T, Garcia de Lomas J, Meyer CU, Bertrand I, Eymin C, Thomas S, Sadorge C. Comparison of intramuscular and subcutaneous administration of a herpes zoster live-attenuated vaccine in adults aged >/=50 years: a randomised non-inferiority clinical trial. Vaccine. 2015 Feb 4;33(6):789-95. doi: 10.1016/j.vaccine.2014.12.024. Epub 2014 Dec 30. PMID 25555381
- [Background] Pinchinat S, Cebrian-Cuenca AM, Bricout H, Johnson RW. Similar herpes zoster incidence across Europe: results from a systematic literature review. BMC Infect Dis. 2013 Apr 10;13:170. doi: 10.1186/1471-2334-13-170. PMID 23574765
- [Background] Nardone A, de Ory F, Carton M, Cohen D, van Damme P, Davidkin I, Rota MC, de Melker H, Mossong J, Slacikova M, Tischer A, Andrews N, Berbers G, Gabutti G, Gay N, Jones L, Jokinen S, Kafatos G, de Aragon MV, Schneider F, Smetana Z, Vargova B, Vranckx R, Miller E. The comparative sero-epidemiology of varicella zoster virus in 11 countries in the European region. Vaccine. 2007 Nov 7;25(45):7866-72. doi: 10.1016/j.vaccine.2007.07.036. Epub 2007 Aug 8. PMID 17919788
- [Background] Calabro GE, Tognetto A, Carini E, Mancinelli S, Sarnari L, Colamesta V, Ricciardi W, de Waure C. Strategies to Improve Vaccination among At-Risk Adults and the Elderly in Italy. Vaccines (Basel). 2020 Jul 4;8(3):358. doi: 10.3390/vaccines8030358. PMID 32635467
- [Background] Valente N, Cocchio S, Stefanati A, Baldovin T, Martinelli D, Prato R, Baldo V, Gabutti G. Temporal trends in herpes zoster-related hospitalizations in Italy, 2001-2013: differences between regions that have or have not implemented varicella vaccination. Aging Clin Exp Res. 2017 Aug;29(4):771-779. doi: 10.1007/s40520-017-0782-z. Epub 2017 Jun 12. PMID 28608255
- [Background] Tartari F, Spadotto A, Zengarini C, Zanoni R, Guglielmo A, Adorno A, Valzania C, Pileri A. Herpes zoster in COVID-19-positive patients. Int J Dermatol. 2020 Aug;59(8):1028-1029. doi: 10.1111/ijd.15001. Epub 2020 Jun 12. No abstract available. PMID 32530063
- [Background] Thomas SL, Hall AJ. What does epidemiology tell us about risk factors for herpes zoster? Lancet Infect Dis. 2004 Jan;4(1):26-33. doi: 10.1016/s1473-3099(03)00857-0. PMID 14720565
- [Background] Esteban-Vasallo MD, Dominguez-Berjon MF, Gil-Prieto R, Astray-Mochales J, Gil de Miguel A. Sociodemographic characteristics and chronic medical conditions as risk factors for herpes zoster: a population-based study from primary care in Madrid (Spain). Hum Vaccin Immunother. 2014;10(6):1650-60. doi: 10.4161/hv.28620. Epub 2014 May 7. PMID 24805130
- [Background] Nimmo A, Steenkamp R, Ravanan R, Taylor D. Do routine hospital data accurately record comorbidity in advanced kidney disease populations? A record linkage cohort study. BMC Nephrol. 2021 Mar 17;22(1):95. doi: 10.1186/s12882-021-02301-5. PMID 33731041
- [Background] Humphries KH, Rankin JM, Carere RG, Buller CE, Kiely FM, Spinelli JJ. Co-morbidity data in outcomes research: are clinical data derived from administrative databases a reliable alternative to chart review? J Clin Epidemiol. 2000 Apr;53(4):343-9. doi: 10.1016/s0895-4356(99)00188-2. PMID 10785564
- [Background] Kim YJ, Lee CN, Lee MS, Lee JH, Lee JY, Han K, Park YM. Recurrence Rate of Herpes Zoster and Its Risk Factors: a Population-based Cohort Study. J Korean Med Sci. 2018 Dec 20;34(2):e1. doi: 10.3346/jkms.2019.34.e1. eCollection 2019 Jan 14. PMID 30636941
- [Background] Fiasca F, Necozione S, Fabiani L, Mastrodomenico M, Mattei A. Measles-Related Hospitalizations in Italy, 2004-2016: The Importance of High Vaccination Coverage. Ann Glob Health. 2019 Mar 19;85(1):40. doi: 10.5334/aogh.2455. PMID 30896136